CLINICAL TRIAL: NCT04721184
Title: Impact of Body Composition on the Prognosis and Toxicity of Patients Diagnosed With Recurrence or Metastasic Squamous Cell Carcinoma of the Head and Neck (SCCHN) Treated With Immune Checkpoint Inhibitors (ICI)
Brief Title: Impact of Low Muscle Mass in HNC Treated With Immunotherapy
Acronym: IMMUNONUTRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Other Study IDs: PR299/20
Record Dates: First submitted 2020-11-25; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Small Cell Carcinoma; Sarcopenia
Keywords: head and neck cancer; immune checkpoint inhibitors; muscle mass; sarcopenia
MeSH Terms: conditions — Sarcopenia; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to evaluate the baseline muscle mass as a predictive biomarker of treatment response in patients with recurrence or metastatic squamous cell carcinoma of the head and the neck (SCCHN) treated with immune checkpoint inhibitors (ICI)

DETAILED DESCRIPTION:
Body composition including sarcopenia (loss of muscle mass), sarcopenic obesity, and mioesteaosis has been well reported to be an independent predictors of mortality, toxicity, and complications in cancer patients with different locations and treatments. However, there are currently no data on impact of body composition and the oncological outcomes in SCCHN patients treated with immune checkpoint inhibitors (ICI) due to recurrence or metastasic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with recurrence or metastatic SCCHN treated with antiPDL1, antiPD1 or antiCTLA-4 drugs, alone or in combination within our institution.
* Patients who have previously signed informed consent.
* Patients with measurable tumor lesions.

Exclusion Criteria:

* Patients with non-measurable lesions.
* Patients who do not sign the informed consent.
* Patients not treated with immunotherapy.
* Patients in a double-blind trial in whom the assigned branch is not known.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A longitudinal prospective study will be carried out of 120 patients with a diagnosis of recurrence or metastatic SCCHN who start treatment with immunotherapy-based regimens at the Institut Català d'Oncologia- L'Hospitalet from November 2020 until the necessary sample size is completed.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the baseline muscle mass as a predictive biomarker of treatment response in patients with recurrence or metastatic squamous cell carcinoma of the head and the neck (SCCHN) treated with immune checkpoint inhibitors (ICI) | at baseline
  Assessed by CT scan at L3 level

SECONDARY OUTCOMES:
- To evaluate the impact of malnutrition and weight loss on overall survival, recurrence-free survival, locoregional control, and toxicity in patients with recurrence or metastatic SCCHN treated with immunotherapy-based regimens. | 2-3 months and 6 months
  Evaluated by full nutritional assessment
Evaluate baseline muscle mass as a predictive biomarker of toxicity | 2-3 months and 6 months
  Assessed by CT scan at L3 level
Evaluate the impact of adipose tissue as a predictor of survival and toxicity | 6 months
  Assessed by CT scan at L3 level including total adipose tissue, subcutaneous, visceral and intramuscular fat mass
Evaluate changes in body composition | 2-3 months and 6 months
  Assessed by CT scan at L3 level
Evaluate the need for nutritional support throughout the treatment and the type if so | through study completion, on average of 6 months
  Evaluated after performed full nutritional assessment by a checklist with all different options
Observe the correlation of a lower muscle mass with an increase in inflammatory parameters and oncological outcomes | 2-3 months and 6 months
  Assessed by CT scan at L3 level and blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Arribas, Principal Investigator — Institut Catlà d'Oncologia
Locations (1):
- Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain